CLINICAL TRIAL: NCT04782739
Title: Evaluation of the Impact of the COVID-19 Pandemic on Provision and Uptake of Services for the Prevention of Mother-to-child Transmission of HIV and Syphilis in Zimbabwe
Brief Title: Impact of COVID-19 on Provision and Uptake of Prevention of Mother-to-child Transmission of HIV Services in Zimbabwe
Status: Completed | Type: Observational
Sponsor: University of Zimbabwe (Other)
Collaborators: Ministry of Health and Child Welfare, Zimbabwe (Other); Centre for Sexual Health and HIV/AIDS Research Zimbabwe (CeSHHAR Zimbabwe) (Other); PENTA Foundation (Network); ViiV Healthcare (Industry); University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: MRCZ/A/2682
Record Dates: First submitted 2021-02-23; First posted 2021-03-04 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections; Syphilis
Keywords: HIV; Syphilis; Pregnancy; Infants; Vertical Transmission; COVID-19
MeSH Terms: conditions — HIV Infections; Syphilis; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Description of PMTCT service provision and uptake at healthcare facilities: Aggregated data will be collected from all 1560 public healthcare facilities in Zimbabwe on key indicators including antenatal testing and treatment of HIV and syphilis, and management of HIV-exposed and HIV-positive infants. Data will be collected from March 2015 (5 years prior to the pandemic) to the end of the study, to explore trends over time.
  Interventions: Other: None - Descriptive study
- Neonatal admissions at Harare Children's Hospital: Individual-level patient data will be collected on all neonates admitted for care at Harare Children's Hospital, including on patient characteristics, clinical status at presentation and outcomes. Data will be collected from February 2019 to the end of the study, to explore trends over time.
  Interventions: Other: None - Descriptive study
- Qualitative study: Qualitative study of 20 pregnant/lactating women accessing routine PMTCT services and 10 community healthcare workers from the Mabvuku and Kuwadzana Polyclinics. The estimated enrolment of 30 participants given in the study design section above refers to participants from this group only.
  Interventions: Other: None - Descriptive study

INTERVENTIONS:
Other: None - Descriptive study — Descriptive study

SUMMARY:
The COVID-19 pandemic and response are likely to lead to severe unintended consequences for the prevention of mother-to-child transmission (PMTCT) of HIV and syphilis. Zimbabwe has made huge progress in coverage of antenatal testing of HIV and syphilis, which reached 98% and 91% in 2019, and is aiming for dual elimination. However, there is emerging evidence of disruption to health services due to COVID-19, similar to that seen in prior epidemics, which may reverse this progress. Mathematical modelling has estimated 3 and 6 month interruptions to ART supply would lead to 1.67 and 2.07 times more babies being born with HIV in SSA over the next year respectively. This study aims to provide real-world data to understand the effects of COVID-19 on the provision and uptake of PMTCT services. Our study has five objectives. Firstly, to conduct a retrospective analysis of national data routinely collected by healthcare facilities to explore changes before, during and after the pandemic in key indicators related to antenatal testing and treatment of HIV and syphilis, and management of HIV-exposed and infected infants. Secondly, data on neonates admitted to Sally Mugabe Central Hospital, already collected for the NeoTree study, will be analysed to explore the impact of COVID-19 on the number of HIV-exposed infants hospitalised, their clinical status at presentation and outcomes. Thirdly, qualitative studies with mothers and healthcare workers will explore barriers to optimal engagement with care and provision of PMTCT services respectively. Fourthly, quantitative results on testing and ART provision will be used to model the impact of disruptions on the rate of PMTCT of HIV enabling policy makers to plan for subsequent waves of COVID-19 and future epidemics. Finally, educational materials will be developed, piloted and disseminated during the project to provide information to pregnant women on safe access to PMTCT services.

DETAILED DESCRIPTION:
Objectives (i) and (ii) will be met by a retrospective analysis of existing MoHCC data sources, allowing a comprehensive description and evaluation of the effects of the pandemic nationally on pMTCT services and, at a local level, on specialised neonatal care. All public healthcare facilities in Zimbabwe complete monthly returns of aggregate data on numbers of women attending antenatal care (ANC) and having HIV and syphilis testing and treatment during pregnancy, and information on HIV testing, prophylaxis for HIV-exposed infants and treatment of HIV-infected infants. These data are entered onto the DHIS-2 platform. Additionally, the national laboratory database includes data on infant HIV PCR testing.

Data will be extracted from the MoHCC DHIS-2 platform for the 5 years prior to measures taken for lockdown for COVID-19 (which started before any significant community transmission of COVID-19), until at least 6 months after the pandemic in Zimbabwe and corresponding measures end (if possible, depending on the course of the pandemic). National data include returns for 1560 healthcare facilities across 10 provinces. Descriptive analyses will focus on the year prior to lockdown, the period of the pandemic/associated response in Zimbabwe and a minimum of 6 months afterwards; we will describe changes in indicators nationally and by province. The national laboratory data will be used as an independent (unlinked) data source to verify trends in EID. Coverage of ART during pregnancy, infant prophylaxis and ART in infants with HIV will be estimated by combining data from MoHCC returns with Spectrum estimates, as is done routinely. Interrupted time series models will be used to estimate trends in indicators across the three time periods (five years pre-pandemic, during the pandemic, 6-months post pandemic), accounting for seasonal patterns and trends prior to the pandemic.

Objective (ii) will be addressed by analysis of NeoTree data. NeoTree is an application used in the neonatal unit at Harare Children's Hospital which combines data collection by healthcare workers in real-time with interactive decision support and education for improving quality of care.

Objective (iii) will use a qualitative design to provide complementary data to enhance the quantitative results. Longitudinal in-depth individual interviews with pregnant and lactating women, and with healthcare workers will be conducted at the Harare. Participants willing and able to provide informed consent will be purposively recruited from the Family and Child Health unit at Harare Children's Hospital. Participants will take part in two waves of data collection, at study start and after six months.

Objective (v) will draw out key messages from this mixed-methods approach for communication and education. We will design, produce and disseminate educational materials in various media. We will build on existing materials already available in Shona (www.picturinghealth.org) and study findings from objectives (i)-(iv) to develop, pilot and evaluate educational materials for women and families on accessing healthcare safely, and disseminate materials to healthcare workers and policymakers. These will include social media targeted video and short animations in Shona, designed to be easily adaptable to other settings for wider dissemination.

ELIGIBILITY:
Group 1:

Inclusion criteria:

• Anonymous aggregated data will be collated retrospectively for all pregnant women/infants receiving care at all public healthcare facilities in Zimbabwe, from March 2015 to the end of the study

Exclusion criteria:

None

Group 2:

Inclusion criteria:

• All neonates admitted to Sally Mugabe Central Hospital, from February 2019 to the end of the study

Exclusion criteria:

None

Group 3 - Pregnant/lactating women:

Inclusion criteria:

* Accessing antenatal or postnatal services at Mabvuku and Kuwadzana clinics
* Have lived in the Mabvuku and Kuwadzana clinics catchment area during the national lockdown
* Willing and able to give written or audio informed consent for participation.
* Willing to participate in the follow-up study

Exclusion criteria:

None

Group 3 - Community healthcare workers

Inclusion criteria:

* Working and interacting directly with women seeking antenatal or postnatal care services
* Working at the health facility/ community during and prior to the lockdown
* Willing and able to give written or audio informed consent for participation.

Exclusion criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group 1:
  Anonymous aggregated data will be collated retrospectively for all pregnant women/infants receiving care at all public healthcare facilities in Zimbabwe, from March 2015 to the end of the study
  Group 2:
  All neonates admitted to Sally Mugabe Central Hospital, from February 2019 to the end of the study
  Group 3:
  Pregnant/lactating women and community healthcare workers from the Mabvuku and Kuwadzana Polyclinics
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of pregnant women seen in antenatal care who are tested for HIV and syphilis | Up to 6 years
  Based on data from Group 1
Proportion of HIV-positive pregnant women seen in antenatal care who are on antiretroviral therapy | Up to 6 years
  Based on data from Group 1
Proportion of HIV-exposed infants seen in antenatal care who are tested for HIV by 6 weeks of age | Up to 6 years
  Based on data from Group 1
Number of HIV-exposed neonates admitted to Sally Mugabe Central Hospital | Up to 2 years
  Based on data from Group 2
Among neonates admitted to Sally Mugabe Central Hospital, number receiving HIV testing and prophylaxis | Up to 2 years
  Based on data from Group 2
Case fatality rate per 1,000 HIV-exposed neonates admitted to Sally Mugabe Central Hospital | Up to 2 years
  Based on data from Group 2
Number of pregnant women who experienced interruptions to PMTCT service delivery | Up to 18 months
  Based on data from Group 3
Qualitative evaluation of the impact of COVID-19 on provision and uptake of PMTCT services | Up to 18 months
  Based on data from Group 3

CONTACTS AND LOCATIONS:
Overall Officials: Mutsa Bwakura-Dangarembizi, Principal Investigator — University of Zimbabwe Clinical Research Centre
Locations (2):
- Zimbabwe (2):
  - Kuwadzana Polyclinic, Harare
  - Mabvuku Polyclinic, Harare

REFERENCES:
- [Result] Chappell E, Chimwaza A, Manika N, Wedderburn CJ, Mupambireyi Nenguke Z, Gannon H, Cowan F, Gibb T, Heys M, Fitzgerald F, Phillips A, Chimhuya S, Gibb DM, Ford D, Mushavi A, Bwakura-Dangarembizi M. Impact of the COVID-19 pandemic on the provision and uptake of services for the prevention of mother-to-child transmission of HIV in Zimbabwe. PLOS Glob Public Health. 2023 Aug 14;3(8):e0002296. doi: 10.1371/journal.pgph.0002296. eCollection 2023. PMID 37578953
- [Result] Gannon H, Chappell E, Ford D, Gibb DM, Chimwaza A, Manika N, Wedderburn CJ, Nenguke ZM, Cowan FM, Gibb T, Phillips A, Mushavi A, Fitzgerald F, Heys M, Chimhuya S, Bwakura-Dangarembizi M. Effects of the COVID-19 pandemic on the outcomes of HIV-exposed neonates: a Zimbabwean tertiary hospital experience. BMC Pediatr. 2024 Jan 5;24(1):16. doi: 10.1186/s12887-023-04473-5. PMID 38183019
- [Result] Mupambireyi Z, Cowan FM, Chappell E, Chimwaza A, Manika N, Wedderburn CJ, Gannon H, Gibb T, Heys M, Fitzgerald F, Chimhuya S, Gibb D, Ford D, Mushavi A, Bwakura-Dangarembizi M. "Getting pregnant during COVID-19 was a big risk because getting help from the clinic was not easy": COVID-19 experiences of women and healthcare providers in Harare, Zimbabwe. PLOS Glob Public Health. 2024 Jan 8;4(1):e0002317. doi: 10.1371/journal.pgph.0002317. eCollection 2024. PMID 38190418